CLINICAL TRIAL: NCT01336699
Title: Safety and Immunogenicity of Two Live, Attenuated Oral Shigella Sonnei Vaccines: WRSs2 and WRSs3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09-0009; HHSN272201300016I
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2015-10-14

CONDITIONS: Shigella Infection
Keywords: Shigella sonnei; shigellosis; vaccine; WRSs2; WRSs3
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort A (Experimental): WRSs2 vaccine 1x10^3 colony-forming units (cfu) orally (8 patients), WRSs3 vaccine 1x10^3 cfu orally (8 patients), Placebo 30 ml orally (2 patients)
  Interventions: Other: Placebo; Biological: WRSs2; Biological: WRSs3
- Cohort B (Experimental): WRSs2 vaccine 1x10^4 colony-forming units (cfu) orally (8 patients), WRSs3 vaccine 1x10^4 cfu orally (8 patients), Placebo 30 ml orally (2 patients)
  Interventions: Other: Placebo; Biological: WRSs2; Biological: WRSs3
- Cohort C (Experimental): WRSs2 vaccine 1x10^5 colony-forming units (cfu) orally (8 patients), WRSs3 vaccine 1x10^5 cfu orally (8 patients), Placebo 30 ml orally (2 patients)
  Interventions: Other: Placebo; Biological: WRSs2; Biological: WRSs3
- Cohort D (Experimental): WRSs2 vaccine 1x10^6 colony-forming units (cfu) orally (8 patients), WRSs3 vaccine 1x10^6 cfu orally (8 patients), Placebo 30 ml orally (2 patients)
  Interventions: Other: Placebo; Biological: WRSs2; Biological: WRSs3
- Cohort E (Experimental): WRSs2 vaccine 1x10^7 colony-forming units (cfu) orally (8 patients), WRSs3 vaccine 1x10^7 cfu orally (8 patients), Placebo 30 ml orally (2 patients)
  Interventions: Other: Placebo; Biological: WRSs2; Biological: WRSs3

INTERVENTIONS:
Other: Placebo — Placebo comparator: 1 or 1.5 ml of sterile normal saline 0.9% added to 30 mL of 0.9% sterile normal saline, given orally.
Biological: WRSs2 — WRSs2 is a live, attenuated Shigella sonnei vaccine product, given orally at five escalating doses from 1x10^3 colony-forming units (cfu) to 1x10^7 cfu.
Biological: WRSs3 — WRSs3 is a live, attenuated Shigella sonnei vaccine product, given orally at five escalating doses from 1x10^3 colony-forming units (cfu) to 1x10^7 cfu.

SUMMARY:
Phase 1, randomized, double-blind, placebo controlled, dose-escalation, inpatient study of single doses of S. sonnei. Health adult subjects, ranging in age from 18 to 45 years of age (inclusive) will be screened. Enroll serial groups up to 90 subjects. The primary objective is to evaluate safety and tolerance of WRSs2 by monitoring presence, frequency and severity of clinical signs and symptoms. A secondary objective is to evaluate the immune response in blood and stool following ingestion of WRSs2 and WRSs3.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo controlled, dose-escalation, inpatient study. Subjects will receive a single oral dose of WRSs2, WRSs3 or placebo. Five doses of each vaccine, ranging from 1x10^3 to 1x10^7 colony forming units (cfu) will be evaluated in this study. For each dose, a cohort of 18 subjects (n=18) will be randomized into 3 groups to receive WRSs2 (n=8), WRSs3 (n=8) and placebo (n=2). The three groups will receive approximately the same inoculum dose. Ingestion of the vaccine will be preceded by ingestion of a sodium bicarbonate buffer. Subjects will be enrolled in serial groups at escalating doses to enable the identification of the dose that minimizes reactogenicity while inducing a robust immune response while allowing for a head-to-head comparison of the 2 vaccine candidates. Dose escalation will proceed by approximately 1 log10 cfu levels based on the observations from the preceding group (up to a maximum dose of 1x10^7 cfu). During the 10-13 day inpatient monitoring period, subjects will be evaluated at least twice daily. This assessment will include asking about any symptoms they may be experiencing, with targeted questions for reactogenic symptoms twice each day. Additional assessments will include daily measurement of vital signs, daily-history directed physical examinations and the collection, and grading (for consistency) of each stool along and weighing of all loose or watery stools. Stool specimens or rectal swabs (if unable to produce a stool) will also be evaluated for grossly visible and occult blood and will be cultured for the presence of the vaccine strain. All volunteers will receive antibiotic therapy 8 days after inoculation (unless meeting criteria for early treatment). Subjects will be discharged after initiating antibiotic treatment and passing 2 consecutive stools (at least 6 hours apart) negative for S. sonnei using standard stool culture and identification techniques. Following evaluation and history-directed physical examination, subjects will be discharged, with follow-up on study days 14+/-1, 28+/-2 and 56+/-4 to provide additional specimens for safety checks or immunology monitoring. Subjects will be given an ice-pack and cooler for collection of a stool sample at home which is to be brought to the clinic on the day of the follow-up visit. An interim safety report will compile findings from the preceding group with the PI's interpretation and plan to go forward. The Data Safety Monitoring board (DSMB)/Safety Monitoring Committee (SMC) or its equivalent must concur with the plan before proceeding. The decision to advance to the next highest dose level will be based solely on the safety profile at the tested dose level and will be made independently for each vaccine candidate. The next inpatient group (at the next higher dose) will not be admitted until a minimum of 4 weeks have elapsed from the time of the preceding group's vaccination to ensure adequate time for safety monitoring. The primary objectives are: to evaluate the safety and clinical tolerance of WRSs2 and WRSs3 by monitoring the presence and severity of clinical signs and symptoms. The secondary objectives are: to evaluate the immune response in blood and stool following ingestion of WRSs2 and WRSs3; to assess frequency and duration of fecal shedding of WRSs2 and WRSs3 following ingestion; and to assess any secondary infectious spread of different vaccine strains (WRSs2 or WRSs3) to subjects.

ELIGIBILITY:
Inclusion Criteria:

- Male or non-pregnant female between 18 and 45 years of age (inclusive). - General good health, without (a) significant medical illness, (b) clinically significant physical examination findings as determined by the PI, and (c) screening laboratory values outside the site's normal limits. - Demonstrate comprehension of the protocol procedures and knowledge of study by passing a written examination (pass grade >/=70 percent) on day -1. - Willing to participate after informed consent obtained. Willingness to participate for an inpatient stay lasting up to 13 days and an outpatient follow-up lasting 6 months from vaccination. Subject must be willing to not smoke during the inpatient stay. - Available for all planned follow-up visits. - Negative serum pregnancy test at screening and negative urine pregnancy test on the day of admission to the inpatient phase for female subjects of childbearing potential. Females of childbearing potential must agree to use an efficacious method of birth control (birth control pills, injection hormonal contraceptive, implant hormonal contraceptive, hormonal patch, IUD, sterilization by hysterectomy or tubal ligation, spermicidal products and barrier methods such as cervical sponge, diaphragm, or condom) within two months of vaccination and during the entire study. Abstinence is acceptable. A woman is eligible if she is monogamous with a vasectomized partner. - Willing to not donate blood for up to 12 months after completion of the inpatient phase of the study - Willing to refrain from participation in another investigational vaccine or drug trial at least until after completion of the 6 month follow-up safety call.

Exclusion Criteria:

- Presence of significant medical conditions such as, gastrointestinal disease (such as active gall bladder disease, peptic ulcer, active gastritis or gastroesophageal reflux disease, inflammatory bowel disease, irritable bowel syndrome, or diverticulitis), or a history of bowel surgery (with an exception of appendectomy, or herniorrhaphy) which in the opinion of the investigator precludes participation in the study. - History of cancer (other than a healed skin lesion), heart disease (in the hospital for a heart attack, have an irregular heartbeat, or have had have postural hypotension in the past year), unconsciousness (other than a single brief "concussion"), seizures (other than with fever when <5 years old), autoimmune disease (trouble fighting off infections), history of arthritis within the past 10 years, or eating disorder. - History within the past 5 years of alcohol or drug abuse, hospitalization for psychiatric illness, history of suicide attempt or confinement for danger to self or others, a diagnosis of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis. Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study. - A positive urine test for opiates. - A chronic disease (such as hypertension, hyperlipidemia or anxiety/depression) for which doses of prescription medications are not stable for at least the past 3 months. - A diagnosis of Diabetes. - Scheduled use of steroids (with the exception of inhaled steroids) or other immunosuppressive medication, medicines to stop diarrhea, or medicines for pain or fever, including non-steroidal anti-inflammatory drugs (i.e. ibuprofen). - History of immunosuppressive illness, or immunodeficiency including IgA deficiency or have household contacts who are immunocompromised. - Screening serological tests positive for HepB, HepC, Human immunodeficiency virus (HIV) or rapid plasma reagin (RPR) (syphilis). - A clinically significant abnormality on physical examination, including a systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg, or a resting pulse >100 beats/min or <55 beats/min (<50 beats/min for conditioned athletes). - Pregnant, nursing, or plan to become pregnant within 6 months of receipt of the study product. - In the 4 weeks following vaccine, subject will be living with or having daily contact with elderly persons aged 70 years or more, diapered individuals, persons with disabilities, children < 5 years old, or a woman known to be pregnant or nursing, or anyone with diminished immunity. This includes contact at home, school, day-care, nursing homes, or similar places. - Are a health care worker, work in a day care center for children or the elderly, or work as food handler. - Work with food, such as in restaurants or cafeterias in the 4 weeks following vaccination. - Have been in the hospital 3 or more times for infections like pneumonia or meningitis, or have known collagen vascular disease (i.e. Systemic Lupus Erythematosus [SLE] or dermatomyositis). - Anti-Shigella sonnei LPS IgG antibody titer in serum >1:2500. - Travel to Shigella endemic area in the past 12 months. - HLA B27 positive during medical screening. - Have abnormal screening llaboratory test results per Table 4 Acceptable Laboratory Values in Section 8.1.2.1 and the clinical laboratory's normal values for complete blood count (CBC) [white blood cells (WBC), Hemoglobin (HgB), platelets, and neutrophil and lymphocyte count], creatinine, total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), s odium, potassium, and urinalysis [urine protein, urine glucose and urine red blood cells (RBC)]. - Stool positive for Salmonella, Shigella, Campylobacter, Cholera or Yersinia, parasites, or pathogenic protozoa. - Allergy to sodium bicarbonate, ciprofloxacin, Bactrim (sulfamethoxazole and trimethoprim), or have a known allergy to any component of the vaccine. - Fewer than 3 stools per week or more than 3 stools per day on a regular basis. Loose or liquid stools other than on an occasional basis. - History of diarrhea in the 2 weeks prior to day of vaccination. - Use of laxatives, antacids, or other agents to lower stomach acidity at least weekly. - History of allergy or intolerance to soy or soy products. - Use of antibiotics during the 7 days before dosing or proton pump inhibitors, H2 blockers, or antacids within 48 hours of dosing. - Have a temperature of >/=100.4 degrees Fahrenheit orally or illness within 3 days of the inpatient visit. - History of or expected exposure to Shigella by infection, challenge, vaccination or laboratory work during the active study period (28 days post vaccination). - Use of any investigational drug or any investigational vaccine within 30 days preceding vaccination, or planned use during the 60 days after receipt of the study agent. - Have taken a licensed, live vaccine within 28 days or a licensed inactivated vaccine within 14 days of receiving this study vaccine. - Long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 ug/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal, intra-articular, and topical steroids are allowed). - Inability to comply with inpatient rules and regulations. - Has any other condition that in the opinion of the Investigator, would jeopardize the safety or rights of a participant or would render the subject unable to comply with the protocol. - Use of prescription and/or over the counter (OTC) medications that contain acetaminophen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs, during the 48 hours prior to investigational product administration. - Receipt of blood or blood products within the past six months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2015-05-12 (Actual); Study Completion 2015-05-12 (Actual)

PRIMARY OUTCOMES:
Frequency, duration, and severity of the following solicited symptoms: diarrhea, nausea, vomiting, fever, and abdominal cramping, also frequency of dysentery, and dehydration, and occurrence of abnormal clinical laboratory values | Day 0-14
Occurrence of vaccine-associated serious adverse events (SAEs) | Day 0 to Day 180

SECONDARY OUTCOMES:
Cell Mediated Immunogenicity: Measure memory B-cell response to Shigella specific antigens. | Day 0, 28 and 56
Fecal shedding of vaccine - duration of detectable fecal presence of WRSs2 and WRSs3 by polymerase chain reaction (PCR) and culture. | Day 0 to 10, 14 and 28
Mucosal immunogenicity: i) IgA-ASC and IgG ASC and ALS response to Shigella antigens: S. sonnei LPS, IpaB, IpaC, IpaD, and S. sonnei Invaplex 50 | Day -1, 5, 7, 9 and 14
Mucosal immunogenicity: ii) Fecal IgA response to Shigella antigens: S. sonnei LPS, IpaB, IpaC, IpaD, and S. sonnei Invaplex 50 | Day -1, 0, 3, 7, 10, 14 and 28
Secondary infectious spread of different vaccine strains to participants. Secondary infections will be measured by assessing fecal shedding using product-specific PCR. | Day 0 to 10, 14 and 28
Systemic immunogenicity: i) Serum IgA, IgM and IgG response to Shigella antigens: S. sonnei Invaplex 50, LPS, IpaB, IpaC, and IpaD | Day -1, 7, 14, 28 and 56

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Venkatesan MM, Ballou C, Barnoy S, McNeal M, El-Khorazaty J, Frenck R, Baqar S. Antibody in Lymphocyte Supernatant (ALS) responses after oral vaccination with live Shigella sonnei vaccine candidates WRSs2 and WRSs3 and correlation with serum antibodies, ASCs, fecal IgA and shedding. PLoS One. 2021 Nov 18;16(11):e0259361. doi: 10.1371/journal.pone.0259361. eCollection 2021. PMID 34793505